CLINICAL TRIAL: NCT06599138
Title: Ultrasound-guided Maxillary Nerve Block: An Anatomical Cadaveric Study. Determination of Dispersion in Ultrasound-guided Suprazygomatic Maxillary Nerve Block in Cadavers.
Brief Title: Maxillary and Mandibular Nerve Block. Block One Get One Free.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Servei Central d'Anestesiologia (Other)
Collaborators: International University of Catalonia (Other)
Responsible Party: Principal Investigator, Gloria Molins Ballabriga, MD, PhD, Servei Central d'Anestesiologia
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: REST-INVI-2024-03
Record Dates: First submitted 2024-06-01; First posted 2024-09-19 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Postoperative Pain; Regional Anesthesia Morbidity
Keywords: Maxillary nerve; Nerve block; Ultrasound
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Injection of 2ml in the pterygopalatine fossa (Other): Perfom an ultrasound-guided maxillary nerve block with injection of 2 ml of contrast in the pterygopalatine fossa
  Interventions: Device: Ultrasound-guided maxillary nerve block
- Injection of 5ml in the pterygopalatine fossa (Other): Perfom an ultrasound-guided maxillary nerve block with injection of 5 ml of contrast in the pterygopalatine fossa
  Interventions: Device: Ultrasound-guided maxillary nerve block

INTERVENTIONS:
Device: Ultrasound-guided maxillary nerve block — Suprazygomatic approach, ultrasound-guided infrazygomatic window, maxillary nerve block for injection of 2 - 5 ml of contrast
  Other Names: Maxillary nerve block

SUMMARY:
Ultrasound-guided maxillary nerve block is mandatory for perioperative pain management of surgeries involving the middle third of the face. The suprazygomatic approach to the maxillary nerve has proven to be the safest and most effective. The volume used for maxillary nerve block remains a matter of debate; and this study aims to compare and study the dispersion of 2 - 5ml injected into the ptergopalatine fossa, and to know the reach of the mandibular nerve with this block.

DETAILED DESCRIPTION:
The second division of the trigeminal nerve, the maxillary nerve (MN), exits the cranial region of the face via the foramen rotundum. From there, it travels laterally and forward through the pterygopalatine fossa, passes through the infra-orbital foramen at the bottom of the pterygomaxillary fossa, and ends up on the floor of the orbit. The MN is a purely sensory nerve that delivers innervation to the lower eyelid, upper lip, cheek, upper dental arch, maxillary sinus, hard and soft palate, posterior nasal cavity, and nasal ala. Effective anesthesia of the maxillary area can be achieved by surgeon's submucosal infiltration, witch appears to change the operative environment, or by inserting a needle in the pterygopalatine fossa (PPF). Although anesthetic infiltration around the mouth cavity or surgical site is simpler to execute than a selective nerve block, it might not be practical in some circumstances, such as when the surgical site is infected or inflamed. Therefore, the maxillary nerve block is preferred over local anesthetic infiltration when the surgical field covers the second third of the face and beyond the oral cavity, for example in maxillary osteotomy. The MN block can also be used for procedures of neurodestruction using neurolytic agents, for permitting anatomic differential neural blockade, and for the diagnostic evaluation of facial pain to determine whether pain is sympathetic or somatic in origin. However, the MN block can result in a number of problems, including as temporal blindness, hematoma formation, diplopia, temporary ophthalmoplegia and ptosis, penetration of the orbit, and brainstem anesthesia. Two approaches for maxillary nerve block in the pterigopalatina fossa have been described: infrazygomatic and suprazygomatic. Several risks associated with the infrazygomatic route of the maxillary block have been described, including the possibility of maxillary artery puncture and orbital or skull penetration. The suprazygomatic approach to maxillary nerve block has been shown to be safer for treating people with trigeminal neuralgia and for the anesthetic management of surgeries of the mid face. The amount of anesthetic injected into the pterygopalatine fossa for MN block is linked to certain issues, whereas other complications are related to the specific anatomical approach used. The typical volume of the PPF in adults has been reported from investigations in dry skulls as close to one ml. However, when executing this block clinically, two to five milliliters are usually injected. As a result, the excess amount of local anesthetic may move intracranially or into the orbit through the infratemporal fossa. Meanwhile, the location of this remaining volume has not been formally investigated.

Due to its many benefits, including safety profile, convenience of use, and low radiation exposure, the use of ultrasound guiding for regional anesthetic and pain mitigation has grown in popularity. Key anatomical features can be identified with its assistance, and by seeing the needle tip as it advances, it facilitates ideal needle insertion. The use of ultrasound pictures has been linked to a variety of superficial to deep nerve blocks in relation to head and neck blocks. Thus, the use of ultrasound for maxillary nerve block for clinical purpose is now mandatory. Although a safe and reliable suprazygomatic MN block technique has been validated providing satisfactory analgesia for midface surgery and chronic maxillofacial pain syndromes, where the remaining local anesthesia diffuses after filling the pterygopalatine fossa in maxillary nerve block has not been formally investigated.

Some authors suggest that with the injection of sufficient volume into the PPF during the maxillary nerve block, some remaining volume could diffuse to the pterygomandibular space, suggesting a communication between the two. And these data could justify the reported high analgesic power of the maxillary nerve block in maxillofacial surgery, which in addition to blocking the branches of the maxillary nerve itself located in the PPF, could also block branches of the mandibular nerve located in the pterygomandibular space. Therefore, randomized controlled trials are needed to determine in greater detail the dispersion of the injected volume outside the PPF when the maxillary nerve block is performed.

The goal of this anatomical study is to identify the extent of local anesthesia spreaded that might influence anesthetic coverage and blockrelated complications.

ELIGIBILITY:
Inclusion Criteria:

- Embalmed cadaveric specimens without known maxillary disease

Exclusion Criteria:

- Embalmed cadaveric specimens with known maxillary disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-11-14 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-16 (Estimated)

PRIMARY OUTCOMES:
Spread of contrast to mandibular nerve branches | 0 hours (After performing the maxillary nerve block)
  To analyze the spread of 2 and 5 ml of injected contrast to branches of the mandibular nerve after suprazygomatic ultrasound-guided single injection into the pterigopalatina fossa.

SECONDARY OUTCOMES:
Spread of contrast to other locations | 0 hours (After performing the maxillary nerve block)
  To analyze the spread of 2 and 5 ml of injected contrast to other locations after suprazygomatic ultrasound-guided single injection into the pterigopalatina fossa.
  Compare different volumes (2 and 5ml) of contrast injected into the pterygopalatine fossa to investigate the location of its dispersion away from the maxillary nerve.

CONTACTS AND LOCATIONS:
Locations (1):
- Anestalia - Servei Central d'Anestesiologia, Barcelona, Spain

REFERENCES:
- [Background] Mesnil M, Dadure C, Captier G, Raux O, Rochette A, Canaud N, Sauter M, Capdevila X. A new approach for peri-operative analgesia of cleft palate repair in infants: the bilateral suprazygomatic maxillary nerve block. Paediatr Anaesth. 2010 Apr;20(4):343-9. doi: 10.1111/j.1460-9592.2010.03262.x. Epub 2010 Feb 23. PMID 20199610
- [Background] Echaniz G, Chan V, Maynes JT, Jozaghi Y, Agur A. Ultrasound-guided maxillary nerve block: an anatomical study using the suprazygomatic approach. Can J Anaesth. 2020 Feb;67(2):186-193. doi: 10.1007/s12630-019-01481-x. Epub 2019 Sep 23. PMID 31549339
- [Background] Kampitak W, Tansatit T, Shibata Y. A Novel Technique of Ultrasound-Guided Selective Mandibular Nerve Block With a Lateral Pterygoid Plate Approach: A Cadaveric Study. Reg Anesth Pain Med. 2018 Oct;43(7):763-767. doi: 10.1097/AAP.0000000000000760. PMID 29659436
- [Background] Poore TE, Carney MT. Maxillary nerve block: a useful technique. J Oral Surg. 1973 Oct;31(10):749-55. No abstract available. PMID 4516663
- [Background] Fujii A. [New technic for blocking the 2nd division of the trigeminal nerve. Experimental and clinical studies on "suprazygomatic route"]. Masui. 1976 Dec;25(13):1370-82. No abstract available. Japanese. PMID 1034732
- [Background] Singh B, Srivastava SK, Dang R. Anatomic considerations in relation to the maxillary nerve block. Reg Anesth Pain Med. 2001 Nov-Dec;26(6):507-11. doi: 10.1053/rapm.2001.26218. PMID 11707787
- [Background] Suresh S, Voronov P. Head and neck blocks in children: an anatomical and procedural review. Paediatr Anaesth. 2006 Sep;16(9):910-8. doi: 10.1111/j.1460-9592.2006.02018.x. PMID 16918651
- [Background] Okuda Y, Takanishi T, Shinohara M, Nagao M, Kitajima T. Use of computed tomography for mandibular nerve block in the treatment of trigeminal neuralgia. Reg Anesth Pain Med. 2001 Jul-Aug;26(4):382. doi: 10.1053/rapm.2001.25059. No abstract available. PMID 11464362
- [Background] Malamed SF, Trieger N. Intraoral maxillary nerve block: an anatomical and clinical study. Anesth Prog. 1983 Mar-Apr;30(2):44-8. No abstract available. PMID 6587797
- [Background] Sved AM, Wong JD, Donkor P, Horan J, Rix L, Curtin J, Vickers R. Complications associated with maxillary nerve block anaesthesia via the greater palatine canal. Aust Dent J. 1992 Oct;37(5):340-5. doi: 10.1111/j.1834-7819.1992.tb00758.x. PMID 1444954
- [Background] Nique TA, Bennett CR. Inadvertent brainstem anesthesia following extraoral trigeminal V2-V3 blocks. Oral Surg Oral Med Oral Pathol. 1981 May;51(5):468-70. doi: 10.1016/0030-4220(81)90002-5. PMID 6941133
- [Background] Stojcev Stajcic L, Gacic B, Popovic N, Stajcic Z. Anatomical study of the pterygopalatine fossa pertinent to the maxillary nerve block at the foramen rotundum. Int J Oral Maxillofac Surg. 2010 May;39(5):493-6. doi: 10.1016/j.ijom.2009.11.002. Epub 2009 Dec 2. PMID 19959336
- [Background] Spinner D, Kirschner JS. Accuracy of ultrasound-guided superficial trigeminal nerve blocks using methylene blue in cadavers. Pain Med. 2012 Nov;13(11):1469-73. doi: 10.1111/j.1526-4637.2012.01480.x. Epub 2012 Oct 8. PMID 23043718
- [Background] Sahar Hafeez N, Sondekoppam RV, Ganapathy S, Armstrong JE, Shimizu M, Johnson M, Merrifield P, Galil KA. Ultrasound-guided greater palatine nerve block: a case series of anatomical descriptions and clinical evaluations. Anesth Analg. 2014 Sep;119(3):726-730. doi: 10.1213/ANE.0000000000000329. PMID 24977913
- [Background] Sola C, Raux O, Savath L, Macq C, Capdevila X, Dadure C. Ultrasound guidance characteristics and efficiency of suprazygomatic maxillary nerve blocks in infants: a descriptive prospective study. Paediatr Anaesth. 2012 Sep;22(9):841-6. doi: 10.1111/j.1460-9592.2012.03861.x. Epub 2012 May 15. PMID 22587691
- [Background] Nader A, Schittek H, Kendall MC. Lateral pterygoid muscle and maxillary artery are key anatomical landmarks for ultrasound-guided trigeminal nerve block. Anesthesiology. 2013 Apr;118(4):957. doi: 10.1097/ALN.0b013e31826d3dfc. No abstract available. PMID 23059449
- [Background] Nader A, Kendall MC, De Oliveria GS, Chen JQ, Vanderby B, Rosenow JM, Bendok BR. Ultrasound-guided trigeminal nerve block via the pterygopalatine fossa: an effective treatment for trigeminal neuralgia and atypical facial pain. Pain Physician. 2013 Sep-Oct;16(5):E537-45. PMID 24077204
- [Background] Nader A, Bendok BR, Prine JJ, Kendall MC. Ultrasound-Guided Pulsed Radiofrequency Application via the Pterygopalatine Fossa: A Practical Approach to Treat Refractory Trigeminal Neuralgia. Pain Physician. 2015 May-Jun;18(3):E411-5. PMID 26000688
- [Background] Kampitak W, Tansatit T, Shibata Y. A Cadaveric Study of Ultrasound-Guided Maxillary Nerve Block Via the Pterygopalatine Fossa: A Novel Technique Using the Lateral Pterygoid Plate Approach. Reg Anesth Pain Med. 2018 Aug;43(6):625-630. doi: 10.1097/AAP.0000000000000790. PMID 29677030

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-16): https://cdn.clinicaltrials.gov/large-docs/38/NCT06599138/Prot_SAP_000.pdf